CLINICAL TRIAL: NCT04798365
Title: Implementation of an Antimicrobial Stewardship Program Targeting Residents With Urinary Tract Infections in Long-term Care Facilities
Brief Title: Antimicrobial Stewardship in UTIs in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 33-035 ex 20/21
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Urinary Tract Infections
Keywords: UTI; antimicrobial stewardship; long term care facility; nursing home
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The main components of the intervention are 1) two sessions of voluntary continuing medical education on the urinary tract infection program in each LTCF for physicians and nursing staff, 2) distribution of educations materials such as written guidelines on antibiotic prescribing including a smart phone friendly version, 3) implementation of the project homepage as a platform to distribute guidelines and educational videos and to enable physicians to ask questions which will be answered by an infectious disease physician.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): No intervention until end of the stuy.

INTERVENTIONS:
Behavioral: Intervention group — medical education and distribution of educations materials
  Arms: Intervention group

SUMMARY:
Background: The widespread inappropriate use of antimicrobial substances drives resistance development at the individual and population level all over the world. In long-term care facilities (LTCF), antibiotics are among the most frequently prescribed medications. More than one third of antibiotics prescribed in LTCFs are for urinary tract infections (UTI). Studies have shown that 30 - 40% of antibiotic courses prescribed in LTCFs were unnecessary and that more than two-thirds were inappropriate based on society guidelines.

Preliminary data: A surveillance study on healthcare-associated UTIs at LTCFs of the Geriatric Health Centers Graz revealed that guideline recommendations on antimicrobial choice were met in only 50% of patients. The most frequently used antimicrobial substances for UTI were quinolones.

Aims: Using a multifaceted bundle of antimicrobial stewardship interventions consisting of clinical practice guidelines, care pathways and local as well as web-based education and training targeting nursing staff as well as physicians we aim to improve the quality of antimicrobial prescriptions for UTIs in four LTCFs in Graz, Austria.

Design: Non-randomized cluster controlled intervention study. Setting: The Geriatric Health Centers Graz are a local institution comprising among others 4 LTCFs (total of 400 beds). These will serve as intervention group. Four LTCFs located in the surroundings of Graz will serve as control group.

Intervention: The main components of the intervention are 1) two sessions of voluntary continuing medical education on the urinary tract infection program in each LTCF for physicians and nursing staff, 2) distribution of educations materials such as written guidelines on antibiotic prescribing including a smart phone friendly version, 3) implementation of the project homepage as a platform to distribute guidelines and educational videos and to enable physicians to ask questions which will be answered by an infectious disease physician.

Outcomes: The primary outcome will be the proportion of adequate prescriptions (adequate in terms of antimicrobial choice). Secondary outcomes include proportion of adequate prescriptions (adequate in terms of decision to treat), number of cases with clinical failure, number of admissions to hospital due to UTI, number of adverse events attributed to antimicrobial treatment for UTI, percentage of extended spectrum betalactamase (ESBL) producing enterobacteria isolated from urinary cultures

ELIGIBILITY:
Inclusion Criteria:

* residents living in the participating long term care facilities who experience urinary tract infections (UTI)

Exclusion Criteria:

* residents without UTI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of adequate prescriptions (adequate in terms of antimicrobial choice) | 2 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Austria (4):
  - Sonnenhof, Fehring
  - Geriatric Health Centres of the City of Graz, Graz
  - Volkshilfe Steiermark, Graz
  - Bezirkspflege-und Seniorenheim Voitsberg, Voitsberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konig E, Kriegl L, Pux C, Uhlmann M, Schippinger W, Avian A, Krause R, Zollner-Schwetz I. Implementation of an antimicrobial stewardship program for urinary tract infections in long-term care facilities: a cluster-controlled intervention study. Antimicrob Resist Infect Control. 2024 Apr 16;13(1):43. doi: 10.1186/s13756-024-01397-2. PMID 38627795